CLINICAL TRIAL: NCT02545166
Title: Validation of a Purine Biosensor in Detecting Acute Cerebral Ischaemia: Carotid Endarterectomy Model in SMARTChip
Acronym: CEMS
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CI163115
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: Stroke; Purines; SMARTChip; Ischaemia; Carotid endarterectomy; Biosensor
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Carotid endarterectomy patients: 40 male and female patients, aged 18 years and over, scheduled for carotid endarterectomy. Fasted pre-operative (arterial and capillary), peri-operative (arterial) and 1-hour and 24-hour post-operative (arterial) blood samples will be collected and analysed for serum purine concentration.
- Control patients: 80 age and sex-matched control patients scheduled for non-vascular, non-oncological day surgery. A single pre-operative fasted capillary (finger-prick) blood sample will be collected and analysed for serum purine concentration.
- Dynamic controls: 10 aortic aneurysm repair patients, 10 critical leg ischaemia patients, 10 endovascular aneurysm repair patients, 10 kidney transplant patients, and 10 free flap surgery patients.
- Local sampling patients: 10 Patients undergoing revascularisation, 10 patients undergoing lower limb surgery with a tourniquet and 5 patients diagnosed with acute compartment syndrome.

SUMMARY:
This study will validate the sensitivity of a purine biosensor (SMARTChip) in detecting acute cerebral ischaemia in a group of patients undergoing elective carotid endarterectomy. The study will also investigate whether blood purine levels are indicative of future risk of stroke by comparing pre-operative blood purine levels in carotid endarterectomy patients (high risk group) and blood purine levels in a group of age and sex-matched controls.

DETAILED DESCRIPTION:
Blood purine levels have been shown to be associated with ischaemic brain conditions. Studies have consistently shown that levels of purines in the blood rise rapidly when oxygen flow to the brain is reduced (hypoxia) and returns to the pre-hypoxic level within 30 minutes upon restoring the oxygen supply. There is therefore the potential for blood purine levels to be used to diagnose strokes more quickly. The investigators have undertaken a programme of work to develop, test and refine a purine biosensor, called SMARTChip. This is a prospective observational study to test the sensitivity of SMARTChip in detecting fluctuations in blood purine levels throughout various stages of carotid endarterectomy. Carotid endarterectomy patients have been chosen for this study because the procedure provides a controlled normoxic and hypoxic brain environment without compromising patient safety and has clear and systematic technical steps which will ensure reliable and robust data. The investigators will test the pre-, peri- and post-operative blood purine levels in 40 patients undergoing carotid endarterectomy at University Hospitals Coventry and Warwickshire NHS Trust, University Hospitals of North Midlands NHS Trust and University Hospitals Birmingham NHS Foundation Trust.

In this study the investigators will also test the hypothesis that purine levels may be predictive of future stroke risk. In a previous study carried out by the trial team patients undergoing carotid endarterectomy, a group that is by definition at increased risk of stroke, were found to have significantly higher purine levels than would be expected in a healthy population. Therefore a case-control study, including 80 patients recruited from the day surgery schedules at the three hospitals as controls and the 40 CEA patients recruited for the observational study as cases, will be undertaken alongside the observational study to assess whether purine levels differ systematically in CEA patients and controls.

ELIGIBILITY:
Inclusion Criteria:

CEA Patients:

* Aged 18 years and over
* Scheduled for carotid endarterectomy

Controls

* Aged 18 years and over
* Scheduled for day surgery

Dynamic controls

* Aged 18 years and over
* Scheduled for open aortic aneurysm repair, critical ischaemic leg surgery (this includes: Femoral endarterectomy, Axillo-Femoral Bypass Graft, Femoral distal bypass, Fem-Fem crossover graft, Axillary bifemoral graft, Aortobifemoral graft, and Femoral popliteal bypass), endovascular aneurysm repair, Kidney transplants, or Free flap surgery.

Local sampling

* Aged 18 and over
* Scheduled for elective lower limb vascular revascularisation, elective lower limb orthopaedic surgery with a tourniquet or diagnosed with acute compartment syndrome requiring a fasciotomy

Exclusion Criteria:

CEA patients:

- Unable/unwilling to provide informed consent

Controls:

* Unable/unwilling to provide informed consent
* History of cerebral ischaemia
* History of cancer
* History of cardiovascular disease
* Unable/unwilling to provide a fasting blood sample

Dynamic controls

* Unable/unwilling to provide informed consent
* History of cerebral ischaemia
* History of cancer (except for Free flap surgery patients)

Local sampling

* Unable/unwilling to provide informed consent
* History of cerebral ischaemia
* History of cancer
* History of cardiovascular disease
* Unable/unwilling to provide a blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 male or female patients, aged 18 years or over, scheduled for carotid endarterectomy and 80 age and sex-matched control patients scheduled for day surgery. 50 dynamic controls. 25 Local sampling patients
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Pre-, peri-, and post-operative arterial serum purine concentration (uM) | 24 hours
  Change in arterial serum purine concentration measured pre-, peri-, and post-operatively in CEA patients

SECONDARY OUTCOMES:
Pre-, and post-operative arterial serum purine concentration (uM) | Baseline
  Arterial serum purine concentration measured pre-operatively in CEA patients, controls and local sampling patients.
Pre-, and post-operative capillary serum purine concentration (uM) | Baseline
  Pre-operative capillary serum purine concentration in CEA patients, controls and local sampling patients.
Local or general anaesthetic | Baseline
  Local or general anaesthetic used during procedure in CEA patients, controls and local sampling patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher HE Imray, MB BS PhD, Study Chair — University Hospitals Coventry and Warwickshire NHS Trust; Jack Fairhead, BM BCh BA, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - University Hospitals Coventry and Warwickshire, Coventry, West Midlands